CLINICAL TRIAL: NCT01241266
Title: China Survey of Peptic Ulcer Bleeding
Acronym: PUB
Status: Completed | Type: Observational
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Other Study IDs: NIS-GCN-DUM-2010/1; D961DL00006
Record Dates: First submitted 2010-11-04; First posted 2010-11-16 (Estimated); Last update posted 2011-12-30 (Estimated); Status verified 2011-12

CONDITIONS: Peptic Ulcer Hemorrhage
Keywords: Peptic Ulcer Bleeding; high risk; None-Interventional Study; he proportion of peptic ulcer bleeding patients who are at high risk (Forrest Ia-IIb)
MeSH Terms: conditions — Peptic Ulcer Hemorrhage

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- 1: Target subject population are the consecutive patients hospitalized due to peptic ulcer bleeding. Subjects should be: ≥18 years; admitted to the hospital with an overt upper GI bleed (hematemesis/coffee ground vomiting, melena, hematochezia and other clin

SUMMARY:
This will be a multicenter prospective observational study carried out in China. The investigators will collect data in a pre-specified Case Report Form. Main data from each patient will include demographics, endoscopy classification, and both endoscopy and pharmacological treatments received by patients. Data from each patient will be prospectively collected from the day the patient is diagnosed as peptic ulcer bleeding by endoscopy and receives endoscopy treatment if the investigator thinks it is needed and up to 30 days afterwards. The proportion of peptic ulcer bleeding patients who are at high risk is the primary outcome variable. High risk is defined as the patients with endoscopy Forrest classification Ia to IIb. The rate and type of endoscopic treatment, the rate of successful endoscopy treatment, the re-bleeding rate and the endoscopic re-treatment rate in high risk peptic ulcer bleeding patients will be collected. The surgery rate and mortality rate in high risk and overall patient population will be calculated.

ELIGIBILITY:
Inclusion Criteria:

* Female and/or male aged 18 years and above
* Admitted to the hospital with an overt upper GI bleeding (hematemesis/coffee ground vomiting, melena, hematochezia and other clinical or laboratory evidence of acute blood loss from the upper GI tract)
* Endoscopy demonstrated peptic ulcer bleeding (Forrest I-III)

Exclusion Criteria:

* If participating in any clinical trial, the subject cannot take part in this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Hospitalized Patients
Sampling Method: Non-Probability Sample
Enrollment: 1044 (Actual)
Dates: Start 2010-11; Primary Completion 2011-07 (Actual); Study Completion 2011-07 (Actual)

PRIMARY OUTCOMES:
The proportion of peptic ulcer bleeding patients who are at high risk (Forrest Ia-IIb). | 1 day

SECONDARY OUTCOMES:
The proportion of peptic ulcer bleeding patients who are at high risk (Forrest Ia-IIb) and receiving endoscopic treatment | 1 day
The proportion of patients receiving endoscopic treatments by type of endoscopic treatmentendoscopic treatment | 5 day
The clinically significant re-bleeding rate of high risk (Forrest Ia-IIb) peptic ulcer bleeding patients treated with or without PPI or H2RA, at 3, 5 and 30 days after successful endoscopy treatment. | 30 days

CONTACTS AND LOCATIONS:
Overall Officials: Karen Atkin, Study Director — Astrazeneca China R&D; Zhaoshen Li, Principal Investigator — Changhai Hospital
Locations (31):
- China (31):
  - Research Site, Hefei, Anhui
  - Research Site, Beijing, Beijing Municipality
  - Research Site, Chongqing, Chongqing Municipality
  - Research Site, Fuzhou, Fujian
  - Research Site, Xiamen, Fujian
  - Research Site, Lanzhou, Gansu
  - Research Site, Guangzhou, Guangdong
  - Research Site, Shenzhen, Guangdong
  - Research Site, Haerbin, Heilongjiang
  - Research Site, Wuhan, Hubei
  - Research Site, Changsha, Hunan
  - Research Site, Jiangyin, Jiangsu
  - Research Site, Nanjing, Jiangsu
  - Research Site, Nantong, Jiangsu
  - Research Site, Nanchang, Jiangxi
  - Research Site, Changchun, Jilin
  - Research Site, Shenyang, Liaoning
  - Research Site, Hohhot, Neimeng
  - Research Site, Jinan, Shandong
  - Research Site, Shanghai, Shanghai Municipality
  - Research Site, Taiyuan, Shanxi
  - Research Site, Xian, Shanxi
  - Research Site, Yangquan, Shanxi
  - Research Site, Chengdu, Sichuan
  - Research Site, Tianjin, Tianjin Municipality
  - Research Site, Ürümqi, Xinjiang
  - Research Site, Kunming, Yunnan
  - Research Site, Fuyang, Zhejiang
  - Research Site, Hangzhou, Zhejiang
  - Research Site, Jinhua, Zhejiang
  - Research Site, Wenzhou, Zhejiang